CLINICAL TRIAL: NCT00755430
Title: Structural and Functional Connectivity in Autism Spectrum Disorders by Using Diffusion Spectrum Imaging and Functional Magnetic Resonance Imaging Studies
Brief Title: Structural and Functional Connectivity in Autism Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 200807036R
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorders (ASD); structural and functional connectivity; diffusion spectrum imaging (DSI); functional magnetic resonance imaging (fMRI); siblings; repeated follow-up measurement
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The subjects will receive blood withdrawal. The blood sample will be used for establishing lymphoblastoid cell lines, which will be used for molecular genetic experiments.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Autism spectrum disorder (ASD) has been given a high priority for genetic and neurobiological study. There is no such information in Asian population and no study has conducted using Diffusion Spectrum Imaging (DSI) to investigate the connectivity throughout the world. Moreover, no follow-up study has been done to examine the developmental changes of structural and functional connectivity. We anticipate to establishing a cohort of 50 ASD and their siblings with complete clinical, neuropsychological, brain imaging, and genetic data for longitudinal study on ASD. Our findings will contribute to our understanding of the structural and functional dysconnectivity for ASD and whether dysconnectivity can be an endophenotype for ASD and used as a biomarker for early diagnosis of ASD.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a pervasive neuro-developmental disorder with prominent reciprocal social and communication impairment and restricted repetitive behavior or interest. Because ASD runs in family, because there is no effective biological treatment, and because early intervention can lead to better outcomes, ASD has been given a high priority for genetic and neurobiological study. Although abnormal brain structure has been reported, there is limited data regarding structural and functional dysconnectivity in autism. There is no such information in Asian population and no study has conducted using Diffusion Spectrum Imaging (DSI) to investigate the connectivity throughout the world. Moreover, no follow-up study has been done to examine the developmental changes of structural and functional connectivity. We thus propose this prospectively follow-up brain imaging study on ASD.

Specific Aims:

1. To investigate the location and extend of structural and functional dysconnectivity and their changes over a 2-year period among children with ASD, as compared to their unaffected siblings and normal controls;
2. To correlate the structural and functional dysconnectivity to clinical severity and neuropsychological functioning;
3. To test the association between brain dysconnectivity and several candidate genes related to the CNS patterning (e.g., RELN, En-2, Wnt, bcl-2); and
4. To test whether neuropsychological and brain imaging findings can be the intermediate phenotype of ASD for genetic studies.

We will recruit 50 children with DSM-IV ASD (autistic disorder and Asperger's disorder) aged 3-15, their siblings, and 50 age-, sex-, and handedness-matached healthy controls. A number of instruments will be used to measure autistic symptoms, functional levels, and cognitive ability (i.e. ADI-R, ADOS, SCQ, SRS, and CAST; WISC-III (WPPSI-R, Bayley), DDST, CPM, and SPM; CPT, WCST, Cambridge Neuropsychological Test Automated Batteries). We will also look directly at the brain for structural and functional connectivity using the DSI and fMRI, respectively. We will repeat the assessments at a 2-year interval. The major tasks consisted of five parts: (1) 3 months-recruitment of subjects, researcher training, and pilot study; (2) 1 years 6 months-clinical, neuropsychological, genetic, DSI and fMRI assessments of 150 subjects; (3) 6 months-data analysis, reports to subjects, and manuscript preparation; (4) 1 years 6 months-same assessment of 150 subjects at a 2-year interval; (5) 4 months-data analysis, reports to subjects, and manuscript preparation.

We anticipate to establishing a cohort of 50 ASD and their siblings with complete clinical, neuropsychological, brain imaging, and genetic data for longitudinal study on ASD. Our findings will contribute to our understanding of the structural and functional dysconnectivity for ASD and whether dysconnectivity can be an endophenotype for ASD and used as a biomarker for early diagnosis of ASD.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the subjects with ASD are:

* that subjects have a clinical diagnosis of autistic disorder, or Asperger disorder defined by the DSM-IV and ICD-10, which was made by a full-time board-certificated child psychiatrist at the first visit and following visits;
* their ages range from 3 to 15 when we conduct the study;
* subjects and their biological parents (and siblings if any) consent to participate in this study for completing clinical and brain imaging assessments and blood withdraw for genetic study (this criteria also applied to the controls).

Exclusion Criteria:

The proband subjects will be excluded from the study if they currently meet criteria or have a history of the following condition as defined by DSM-IV:

* Schizophrenia
* Schizoaffective Disorder
* Organic Psychosis
* severe neurological disease. Moreover, the subjects will also be excluded from the study if they completely cannot cooperate with MRI assessments.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The sample will consist of 50 children with DSM-IV ASD (autistic disorder and Asperger's disorder) aged 3-15, their siblings, and 50 age-, sex-, and handedness-matached healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan